CLINICAL TRIAL: NCT00288262
Title: Melatonin Effects on Luteinizing Hormone
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Scripps Health (Other)
Collaborators: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-101 (Scripps SOPRS #); NIH M01 RR00833 (in part)
Record Dates: First submitted 2006-01-30; First posted 2006-02-07 (Estimated); Last update posted 2006-02-07 (Estimated); Status verified 2005-10

CONDITIONS: Hot Flashes
Keywords: hot flashes; melatonin; depression; sleep; luteinizing hormone; postmenopause
MeSH Terms: conditions — Hot Flashes; Depression | interventions — Melatonin

INTERVENTIONS:
Drug: melatonin 0.5 mg

SUMMARY:
In many mammals, the duration of the nocturnal melatonin elevation regulates seasonal changes in reproductive hormones such as luteinizing hormone (LH). Melatonin's effects on human reproductive endocrinology are uncertain. It is thought that the same hypothalamic pulse generator may both trigger the pulsatile release of GnRH and LH and also cause hot flashes. Thus, if melatonin suppressed this pulse generator in postmenopausal women, it might moderate hot flashes. This clinical trial tested the hypothesis that melatonin could suppress LH and relieve hot flashes.

DETAILED DESCRIPTION:
Twenty postmenopausal women troubled by hot flashes underwent one week of baseline observation followed by 4 weeks of a randomized controlled trial of melatonin or matched placebo. The three randomized treatments were melatonin 0.5 mg 2.5-3 hours before bedtime, melatonin 0.5 mg upon morning awakening, or placebo capsules. Twelve of the women were admitted to the GCRC at baseline and at the end of randomized treatment for 24-hour sampling of blood for LH. Morning urine samples were collected twice weekly to measure LH excretion. Subjective responses measured throughout baseline and treatment included sleep and hot flash logs, the CESD and QIDS depression self-ratings, and the SAFTEE physical symptom inventory.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman
* Troubled by hot flashes

Exclusion Criteria:

* Use of reproductive hormones other than continuous estrogen or progesterone hormone replacement
* Any acute illness
* Any anticipated changes of medication
* Anemia (hemoglobin <12) or poor veins Recent trans-time-zone jet travel, shift work, or irregular sleep habits Any neurological or pituitary disease

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-06; Study Completion 2005-02

PRIMARY OUTCOMES:
Hot flashes log
Sleep log
QIDS
CESD
Luteinizing hormone (urine)
Luteinizing hormone (blood)

SECONDARY OUTCOMES:
SAFTEE inventory of symptoms and adverse effects
Other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Kripke, MD, Principal Investigator — Scripps Clinic Sleep Center
Locations (1):
- Scripps Clinic Sleep Center, La Jolla, California, United States